CLINICAL TRIAL: NCT00017381
Title: Dose Finding Study of IDEC-Y2B8 With Autologous Stem Cell Support
Brief Title: Monoclonal Antibody Therapy and Peripheral Stem Cell Transplant in Treating Patients With Non-Hodgkin's Lymphoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03156; J0004
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2013-01

CONDITIONS: Contiguous Stage II Adult Diffuse Large Cell Lymphoma; Contiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Contiguous Stage II Grade 1 Follicular Lymphoma; Contiguous Stage II Grade 2 Follicular Lymphoma; Contiguous Stage II Grade 3 Follicular Lymphoma; Contiguous Stage II Mantle Cell Lymphoma; Contiguous Stage II Marginal Zone Lymphoma; Contiguous Stage II Small Lymphocytic Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Noncontiguous Stage II Grade 1 Follicular Lymphoma; Noncontiguous Stage II Grade 2 Follicular Lymphoma; Noncontiguous Stage II Grade 3 Follicular Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Noncontiguous Stage II Marginal Zone Lymphoma; Noncontiguous Stage II Small Lymphocytic Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Stage I Adult Diffuse Large Cell Lymphoma; Stage I Adult Diffuse Small Cleaved Cell Lymphoma; Stage I Grade 1 Follicular Lymphoma; Stage I Grade 2 Follicular Lymphoma; Stage I Grade 3 Follicular Lymphoma; Stage I Mantle Cell Lymphoma; Stage I Marginal Zone Lymphoma; Stage I Small Lymphocytic Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Small Lymphocytic Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Small Lymphocytic Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — Rituximab; Cyclophosphamide; Filgrastim; Granulocyte Colony-Stimulating Factor; ibritumomab tiuxetan; Peripheral Blood Stem Cell Transplantation

ARMS (1):
- Treatment (Experimental): PART I: Patients receive rituximab IV on days 1, 8, 15, and 22 and cyclophosphamide IV over 1 hour on day 25. G-CSF is administered SC daily beginning on day 26 and continuing until autologous PBSC are harvested.
  PART II: Beginning 4-6 weeks after completion of the fourth rituximab infusion, patients receive indium In 111 ibritumomab tiuxetan IV over 10 minutes on day 1 followed by dosimetry imaging on days 1, 2, 4, and 7. Patients then receive IDEC-Y2B8 IV over 10 minutes once between days 8-15.
  PART III: All patients undergo PBSCT beginning after residual bone marrow radioactivity resolves. G-CSF is administered SC beginning 1 day after PBSCT and continuing until blood counts recover.
  Interventions: Biological: rituximab; Drug: cyclophosphamide; Biological: filgrastim; Radiation: yttrium Y 90 ibritumomab tiuxetan; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Biological: filgrastim — Given SC
  Other Names: G-CSF; Neupogen
Radiation: yttrium Y 90 ibritumomab tiuxetan — Given IV
  Other Names: 90Y ibritumomab tiuxetan; IDEC Y2B8; Y90 Zevalin; Y90-labeled ibritumomab tiuxetan
Procedure: peripheral blood stem cell transplantation — Undergo PBSCT
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell

SUMMARY:
This phase I trial is studying how well monoclonal antibody therapy with peripheral stem cell transplant works in treating patients with non-Hodgkin's lymphoma. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Peripheral stem cell transplant may allow the doctor to give higher doses of monoclonal antibodies and kill more cancer cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose of IDEC-Y2B8 when administered with rituximab in vivo purging and autologous stem cell rescue.

II. To obtain correlative laboratory data of in vivo purging with rituximab in patients with 0-35% marrow involvement.

OUTLINE: This is a multicenter, dose-escalation study of yttrium Y 90 ibritumomab tiuxetan (IDEC-Y2B8).

PART I: Patients receive rituximab IV on days 1, 8, 15, and 22 and cyclophosphamide IV over 1 hour on day 25. Filgrastim (G-CSF) is administered subcutaneously (SC) daily beginning on day 26 and continuing until autologous peripheral blood stem cells (PBSC) are harvested.

PART II: Beginning 4-6 weeks after completion of the fourth rituximab infusion, patients receive indium In 111 ibritumomab tiuxetan IV over 10 minutes on day 1 followed by dosimetry imaging on days 1, 2, 4, and 7. Patients then receive IDEC-Y2B8 IV over 10 minutes once between days 8-15.

The initial 3 patients receive the same dose of IDEC-Y2B8 and then subsequent cohorts of 3-5 patients receive escalating doses of IDEC-Y2B8 until the maximum tolerated dose is determined.

PART III: All patients undergo PBSC transplantation (PBSCT) beginning after residual bone marrow radioactivity resolves. G-CSF is administered SC beginning 1 day after PBSCT and continuing until blood counts recover.

Patients are followed every 3 months for 1 year and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a biopsy-proven indolent or diffuse large B-cell non-Hodgkin's lymphoma as defined as REAL classification marginal zone/MALT, mantle cell, plasmacytoid, lymphoplasmacytoid, small lymphocytic lymphoma or follicle center grades I, II, III or diffuse large B-cell (CLL patients will not be eligible); transformation from a low grade to intermediate or high grade lymphoma is also permissible; patients with diffuse large cell lymphoma must not be eligible for any known potentially curative therapy; at least one diagnostic pathologic specimen will be reviewed by the JHH Pathology Department
* Patients must have received at least one but not more than five prior chemotherapy regimens for treatment of their lymphoma
* Patients may not have received prior external beam radiation therapy to > 25% of active bone marrow (involved field or regional)
* Patients must have 0-35% morphologically identifiable tumor in the trabecular space on bone marrow biopsy; in patients with lymphomas in whom tumor is morphologically difficult to distinguish from normal cells, flow cytometry must show 0-35% identifiable tumor within 4 weeks of registration
* Patients must have =< 35% bone marrow involvement with tumor due to risk of engraftment failure
* Patients may not have hypocellular bone marrow (=< 15% cellularity) or marked decrease in any one (or more) hematopoietic precursor
* Patients may not have received prior murine compounds due to risk of HAMA formation
* WBC must be >= 3,000
* Total lymphocyte count must be < 5,000
* Hgb must be >= 10.0
* Platelets must be >= 75,000
* Serum creatinine must not be greater than 2.0 mg/dl
* Direct bilirubin must be =< 2mg/dl unless secondary to tumor
* AST or ALT must be < 2 x the upper limit of normal
* Normal (>= 45%) left ventricular cardiac ejection fraction, (determined by echocardiogram or MUGA scan)
* DLCO must be > 50% predicted
* Patients with active infections requiring oral or intravenous antibiotics are not eligible for entry onto the study until resolution of the infection
* ECOG performance status =< 2
* Not pregnant (confirmed by serum pregnancy test in females of reproductive potential) or breast feeding, because it is unknown what effect these drugs will have on children
* Women of childbearing potential and sexually active males are strongly advised to use an accepted and effective method of contraception
* Patients with a second malignancy other than basal cell carcinoma or squamous cell carcinoma of the skin or in situ carcinoma of the cervix are not eligible unless the tumor was treated with curative intent at least two years previously
* Women and minorities are encouraged to participate
* Patients who have received prior anti-CD20 therapy must have achieved a partial or complete response
* Patients who are HIV positive will be excluded due to increased risk for bone marrow suppression and other toxicities
* Patients who have received prior radioimmunotherapy, for example Zevalin or Bexxar, are not eligible

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2001-04; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
MTD, defined in terms of clinical toxicities graded using the CTC version 2.0 | Up to day 15
  The modified continual reassessment method (CRM) will be employed to estimate the MTD.

CONTACTS AND LOCATIONS:
Overall Officials: Lode Swinnen, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States